CLINICAL TRIAL: NCT04777188
Title: Left Ventricular Systolic Function After Percutaneous Intramyocardial Septal Radiofrequency Ablation for Hypertrophic Obstructive Cardiomyopathy: a Study Focused on Speckle Tracking Echocardiography
Brief Title: Speckle Tracking Echocardiography Analysis of Left Ventricular Myocardium After Percutaneous Intramyocardial Septal Radiofrequency Ablation for Hypertrophic Obstructive Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Liu Liwen, Director, Xijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20162042-1
Record Dates: First submitted 2021-02-03; First posted 2021-03-02 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
Keywords: Cardiomyopathy, hypertrophic; Speckle tracking echocardiography
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypertrophic Obstructive Cardiomyopathy (Experimental): Left ventricular systolic function by speckle tracking echocardiography before and after percutaneous intramyocardial septal radiofrequency ablation for hypertrophic obstructive cardiomyopathy.
  Interventions: Procedure: Percutaneous Intramyocardial Septal Radiofrequency Ablation for hypertrophic obstructive cardiomyopathy

INTERVENTIONS:
Procedure: Percutaneous Intramyocardial Septal Radiofrequency Ablation for hypertrophic obstructive cardiomyopathy — Under transthoracic echocardiography (TTE) guidance, the puncture site is positioned at the apex. A guiding line is applied along the septal long axis and the radiofrequency ablation electrode needle(17G, Cool-tip™ RF Ablation System and Switching Controller;Medtronic, Minneapolis, MN, USA) pierced towards the hypertrophic anterior interventricular septum (AIVS) 8-10 mm from the subaortic valve. Each ablation lasts for up to 12 min and the ablation power is gradually increased from 30-40W. Then, the ablation needle is withdrawn 10 mm to prepare for the next application. Overall, 3-4 applications are performed in each patient. The ablation creates an area of thermal coagulative myocardial necrosis that appears as a hyperechogenic reflection detected by TTE. If deemed necessary, we repeat the procedure at the posterior interventricular septum (PIVS).

SUMMARY:
Objective to investigate the left ventricular (LV) systolic function by speckle tracking echocardiography before and after percutaneous intramyocardial septal radiofrequency ablation for hypertrophic obstructive cardiomyopathy (HOCM).

Percutaneous intramyocardial septal radiofrequency ablation (named Liwen Procedure) is a safe and effective treatment approach for HOCM and results in sustained improvement in exercise capacity and persistent in reducing left ventricle outflow tract (LVOT) gradient. However, the systolic function of the myocardial after Liwen procedure in HOCM patients is not well exploration and research. Strain evaluation using speckle tracking echocardiography is an excellent tool for assessing regional and global LV functions.

In this study, the investigators aimed to characterize regional and global strain using speckle tracking echocardiography to assess LV radial, circumferential and longitudinal systolic myocardial function in patients with HOCM before and after Liwen procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptoms that limit daily activities (New York Heart Association functional class >II, exercise-induced syncope) despite adequate medical treatment or when medical treatment is not tolerated
2. Patients with a peak LVOT gradient≥50 mm Hg

Exclusion Criteria:

1. Those with a peak instantaneous Doppler LVOT gradient of <50 mm Hg
2. Those with an indication for septal reduction therapy and other lesions requiring surgical intervention (e.g., mitral valve repair/replacement and papillary muscle intervention)
3. Those with end-stage heart failure；and those the echocardialology image quality is not clear enough for strain analysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-10-22 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Left ventricular systolic function before and after Percutaneous Intramyocardial Septal Radiofrequency Ablation | 1 year
  The left ventricular(LV) systolic function was analyzed by Tomtec Workstation with related software. LV was automatically divided into 16 segments using standard segmentation. The following LV parameters were automatically calculated by the software. The 3D strain indexes derived included ,LV peak systolic global longitudinal strain (GLS,percent), LV peak systolic global radial strain (GRS,percent), LV peak systolic global circumferential strain (GCS,percent)

SECONDARY OUTCOMES:
left ventricular outflow tract gradient before and after Percutaneous Intramyocardial Septal Radiofrequency Ablation | 1 year
  The results were obtained by continuous Doppler echocardiography (mmHg)
Interventricular septal thickness before and after Percutaneous Intramyocardial Septal Radiofrequency Ablation | 1 year
  The results were obtained by echocardiography , the unit of mm

CONTACTS AND LOCATIONS:
Locations (1):
- Ultrasound Medicine Department of Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Li J, Zhang J, Shi Y, Sievert H, Taub CC, Bertog S, Ta S, Changhui L, Senser E, Wang J, Hu R, Huang J, Ruan F, Han Y, Li X, Wang B, Zhao X, Liu J, Hsi DH, Liu L. Myocardial mechanics of percutaneous intramyocardial septal radiofrequency ablation. Heart. 2023 Jan 27;109(4):289-296. doi: 10.1136/heartjnl-2022-321597. PMID 36270787